CLINICAL TRIAL: NCT01813929
Title: Effect of Metformin on Vascular and Mitochondrial Function in Type 1 Diabetes
Acronym: MeT1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0693
Record Dates: First submitted 2012-09-28; First posted 2013-03-19 (Estimated); Results first posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Insulin; Metformin; Vascular; Vessels; Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Six week intervention: Study drug/placebo will be given in a forced uptitration with 500 mg once daily for one week, 500 mg twice daily for one week, 500/1000 for one week, and then 1000mg twice daily for the remainder of the 6 week intervention. If uptitration is not tolerated, max dose will be max tolerated dose of at least 500 mg twice daily.
  Other Names: glucophage
  Arms: Metformin
Drug: Placebo — Six-week intervention: Study drug/placebo will be given in a forced uptitration with 500 mg once daily for one week, 500 mg twice daily for one week, and then the higher dose (850 mg) for the remainder of the 6 week intervention.
  Arms: Placebo

SUMMARY:
Insulin resistance (IR) is an important contributor to increased cardiovascular disease risk in type 1 diabetes (T1D). The purpose of this study is to measure the effect of metformin on insulin sensitivity, vascular function and compliance, and mitochondrial function in T1D. The long term goal is to identify novel non-glycemic approaches to managing cardiovascular disease risk in T1D. The results of this study may validate a novel approach to T1D treatment that could significantly improve current management of cardiovascular disease risk in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-59 years of age,
* Type 1 diabetes based on antibody-positivity, rapid persistent conversion to insulin requirement after diagnosis, absent C-peptide, or DKA at diagnosis, or a clinical course consistent with T1D,
* HbA1c 6.0 - 9.5, and
* Willing and able to commit to two 6 week-long periods of blinded medication followed by hyperinsulinemic euglycemic clamp, vascular testing, and muscle biopsies.

Exclusion Criteria:

* Any comorbid condition associated with:

  * inflammation,
  * insulin Resistance, or
  * dyslipidemia including:

    1. cancer,
    2. heart failure,
    3. active or end stage liver disease,
    4. kidney disease, or
    5. rheumatological disease;
* Tobacco use;
* Pregnancy or women who are breastfeeding;
* Steroid use;
* Scheduled strenuous physical activity >3 days a week;
* Angina, known CAD, or any other cardiovascular or pulmonary disease;
* A history of COPD or asthma;
* Presence of systolic blood pressure >190 at rest or >250 with exercise, or diastolic pressure >95 at rest or >105 with exercise;
* Untreated thyroid disease;
* Proteinuria (urine protein >200 mg/dl) or a creatinine > 1.5 mg/dl (males) or 1.4 mg/dL (females), suggestive of severe renal disease;
* Severe Proliferative retinopathy;
* Niacin treatment;
* Administration of experimental agent for T1D within 30 days prior to screening;
* Recent (prior 6 months) or current metformin or thiazolidenedione use;
* Hypoglycemia unawareness or recurrent severe hypoglycemia (no symptoms of hypoglycemia with FSBS<40 and episodes of this severity >1 per week);
* Weight instability (weight change >5% in last 6 months);
* History of any organ transplant, including islet cell transplant;
* Current or prior infection with HIV, hepatitis B or hepatitis C or hepatic -insufficiency (AST or ALT > 2x the upper limits of normal);
* Any condition, medical or otherwise that would, in the opinion of the investigator, prevent complete participation in the study, or that would pose a significant hazard to the subject;
* History of substance abuse within the 12 months prior to screening.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-06; Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Schauer, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants screen failed before starting the study. 3 more participants withdrew after randomization, but before starting the study.
Groups:
- Metformin, Then Placebo: Metformin: Six week intervention: Study drug/placebo will be given in a forced uptitration with 500 mg once daily for one week, 500 mg twice daily for one week, 500/1000 for one week, and then 1000mg twice daily for the remainder of the 6 week intervention. If uptitration is not tolerated, max dose will be max tolerated dose of at least 500 mg twice daily.
  Placebo: Six-week intervention: Study drug/placebo will be given in a forced uptitration with 500 mg once daily for one week, 500 mg twice daily for one week, and then the higher dose (850 mg) for the remainder of the 6 week intervention.
- Placebo, Then Metformin: Placebo: Six-week intervention: Study drug/placebo will be given in a forced uptitration with 500 mg once daily for one week, 500 mg twice daily for one week, and then the higher dose (850 mg) for the remainder of the 6 week intervention.
  Metformin: Six week intervention: Study drug/placebo will be given in a forced uptitration with 500 mg once daily for one week, 500 mg twice daily for one week, 500/1000 for one week, and then 1000mg twice daily for the remainder of the 6 week intervention. If uptitration is not tolerated, max dose will be max tolerated dose of at least 500 mg twice daily.
Period: Overall Study
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin
Started | 5 | 12
Completed Intervention 1 | 5 | 12
Completed Washout (2weeks up to 2 Months) | 5 | 11
Started Intervention 2 | 5 | 11
Completed | 5 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline information was collected for all participants for which outcome measure data was able to be collected. One subject only completed the placebo arm and is not included in paired t-tests.
  Initial random order, double-blinded design was revised to placebo-metformin, single-blinded (participants) design due to concern for carryover effects from metformin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin, Then Placebo | Placebo, Then Metformin | Total
Number analyzed (Participants) | 5 | 12 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (14.4) | 43.3 (11.6) | 43.2 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 1 | 7 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 10 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 12 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 12 | 17

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity by Hyperinsulinemic Euglycemic Clamp
Description: Determine the effect of metformin on insulin sensitivity in T1D. Reported measure is glucose infusion rate during hyperinsulinemic euglycemic clamp normalized to total body weight. For this measure, insulin was infused at 40 mU/m2 surface area. Blood sugar wass checked every 5 minutes and glucose infusion adjusted to maintain glucose level at 90 mg/dL for 2 hours. The glucose infusion rate for the final 30 minutes is reported as GIR (aka M-value or glucose disposal rate) in mg glucose/kg*min. A higher value corresponds to greater sensitivity to insulin. There is no strictly defined normal range.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
mg/kg/min | 3.27 (1.51) | 3.46 (2.15)

2. Primary Outcome: Flow-mediated Brachial Artery Dilation
Description: Measure of endothelial function by brachial ultrasound of the percent dilation after 5 minutes of occlusion.
Time Frame: End of each 6 week intervention period
Population: Not completed on last subjects -futility, concern re reliability, and difficulty getting US images analyzed.
Measure: Mean (Standard Deviation); unit: percent change in BA diameter
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 13
percent change in BA diameter | 8.19 (3.85) | 7.45 (5.86)

3. Secondary Outcome: Arterial Stiffness by PWV
Description: Pulse wave velocity by Sphygmacor as a measure of aortic stiffness in m/sec.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 16
m/sec | 8.64 (2.76) | 8.56 (3.02)

4. Secondary Outcome: Arterial Stiffness by AI@75
Description: Augmentation index by Sphygmacor is a measure of aortic arterial stiffness. AI@75 is the ratio of augmented pressure/pulse pressure adjusted to a heart rate of 75.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 17
ratio | 15.89 (9.08) | 14.96 (12.48)

5. Secondary Outcome: Mitochondrial Measures: Oxygen Consumption
Description: Oxygen consumption rate with various substrates and max uncoupled O2 consumption.
  Measure is performed on permeabilized muscle fibers from biopsy tissue from the vastus lateralis using the Oroboros OxygraphO2k high resolution respirometer. State 3 is full coupled oxygen flux using PMG or PMGS (pyruvate, malate, glutamate, +/- succinate) or OCMS (octanyl carnitine, malate, +/- succinate) as substrates. state 4 is after addition of oligomycin to inhibit the ATP synthase and thus corresponds to the maximum leak state where O2 consumption is limited by the buildup of the proton gradient and can only proceed as fast as the protons can leak back across the membrane. FCCP is added as an uncoupler, allowing free leakage of protons across the inner membrane, and thus measures maximum possible O2 flux. There are no defined normal ranges, but higher state 3 and uncoupled flux indicate better mitochondrial function, while state 4 is needed to correct state 3 to the fully coupled flux.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: pmoles/mg/s
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 15 | 15
pmoles/mg/s
  PMG State 3 Oxygen Flux | 28.3 (6.8) | 29.7 (11.0)
  PMGS State 3 Oxygen Flux | 44.3 (16.5) | 41.5 (16.1)
  PMGS State 4 Oxygen Flux | 14.6 (8.0) | 14.0 (6.3)
  PMGS Uncoupled Max Oxygen Flux | 76.0 (26.3) | 76.4 (21.2)
  OCM State 3 Oxygen Flux | 16.8 (7.0) | 18.0 (5.6)
  OCMS State 3 Oxygen Flux | 43.8 (16.9) | 42.8 (13.1)
  OCMS State 4 Oxygen Flux | 14.6 (7.4) | 15.1 (5.9)
  OCMS Uncoupled Max Oxygen Flux | 67.1 (23.3) | 71.3 (18.8)

6. Secondary Outcome: Mitochondrial Measures: Protein Expression Levels of Electron Transport Chain Complexes
Description: Mito content by Western Blotting of electron transport chain complexes I, II, III, and V. complex 1 utilizes NADH from pyruvate/malate/glutamate while complex II utilizes FADH from succinate. complex III is the cytochrome c reductase while complex V is the ATP synthase.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 11 | 11
Arbitrary units
  complex I | 1436 (981) | 1084 (718)
  complex II | 4375 (2022) | 4201 (1541)
  complex III | 10361 (5131) | 9001 (5451)
  complex V | 23118 (9281) | 23254 (8368)

7. Secondary Outcome: Inflammatory Marker: hsCRP
Description: hsCRP (mg/L) by Beckman Coulter assay
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
mg/L | 2.13 (2.29) | 2.95 (2.75)

8. Secondary Outcome: Heart Rate Variability
Description: measure of autonomic function: ratio of fastest to slowest heart rate during valsalva maneuver
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
ratio | 1.55 (0.34) | 1.42 (0.18)

9. Secondary Outcome: Continuous Glucose Monitor Measures of Mean Glucose
Description: Mean Glucose & Glucose Standard Deviation (Glycemic Variability) by Dexcom CGM
Time Frame: Last Week of each 6 Week Intervention Period (over 7 days)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 14 | 17
mg/dL
  Mean 7 Day Glucose | 162 (35) | 163 (26)
  Glucose Standard Deviation (variability in glucoses throughout the 7 day period) | 64 (14) | 68 (21)

10. Secondary Outcome: Continuous Glucose Monitor Measures of Hypoglycemia
Description: Percent of time less than 70 mg/dL during the final week of each phase by Dexcom CGM.
Time Frame: Last Week of each 6 Week Intervention Period (over 7 days)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 14 | 17
percentage of time | 8.4 (10.7) | 7.9 (6.9)

11. Secondary Outcome: Metabolic Markers: Glucagon
Description: Glucagon (pg/ml); baseline on AM of each phase final study visit.
Time Frame: End of each 6 week intervention period
Population: NS by paired t-test
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
pg/ml | 95.5 (27.8) | 90.2 (45.6)

12. Secondary Outcome: Metabolic Markers: Glucose, Triglycerides, Cholesterol
Description: Glucose (mg/dL), triglycerides (mg/dL), cholesterol (mg/dL) at baseline after each phase
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
mg/dL
  Glucose | 135 (45) | 124 (46)
  Triglycerides | 98 (50) | 78 (41)
  total cholesterol | 156 (38) | 154 (48)

13. Secondary Outcome: Metabolic Markers: Fatty Acids
Description: fatty acids (microeq/L) at baseline after each phase in the AM of the final visit
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: microEq/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
microEq/L | 531 (174) | 446 (185)

14. Secondary Outcome: Metabolic Markers: Glycerol
Description: glycerol (micromol/L) at baseline after each phase in the AM of the final phase visit
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: microM/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
microM/L | 95 (33) | 87 (31)

15. Secondary Outcome: Metabolic Markers: Insulin
Description: insulin (microIU/ml) at baseline after each phase in the AM of the final phase visit
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: microIU/ml
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
microIU/ml | 33.9 (34.3) | 49.1 (56.8)

16. Secondary Outcome: Metabolic Markers: Lactate
Description: lactate (mmol/L) at baseline after each phase in the AM of the final phase visit
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: mmoles/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
mmoles/L | 0.79 (0.26) | 0.75 (0.2)

17. Secondary Outcome: Metabolic Markers: Adiponection
Description: adiponection (microg/ml) at baseline after each phase in the AM of the final phase visit
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: microg/mL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
microg/mL | 13.5 (8.1) | 15.1 (9.4)

18. Secondary Outcome: Vascular Markers: Endothelin-1 (pg/ml)
Description: endothelin-1 at baseline after each phase in the AM of the final phase visit by peninsula labs radioimmunoassay
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 13 | 14
pg/mL | 6.3 (4.8) | 5.8 (2.1)

19. Secondary Outcome: In Vivo Mitochondrial Function: Ratio of the Amount of ATP Generated Per Unit of Oxygen Consumed
Description: Measured by 31P-mass spec. This ratio measures mitochondrial efficiency. The higher the ratio, the more efficiently the individual converts metabolic substrates into ATP, with the ATP then available for energy-demanding cellular processes such as protein synthesis and biomass production
Time Frame: End of each 6 week intervention period
Population: 2 subjects complete data for metformin, but not placebo. (images not good) ME not reported for one placebo subject due to AnGly out of range.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 11 | 8
ratio | 0.152 (0.067) | 0.116 (0.044)

20. Secondary Outcome: In Vivo Mitochondrial Function: Time Constants
Description: Measured by 31P-mass spec. ADP time constant and phosphocreatine time constant. ADP time constant is a measure of the time required to convert ADP → ATP and is a measure of muscle mitochondrial health (energy metabolism). A faster recovery is a better outcome; a slower recovery is a worse outcome. Similarly for phosphocreatine.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 11 | 9
seconds
  ADP time constant | 18.4 (5.4) | 23.3 (10.3)
  Phosphocreatine time constant | 32.9 (9.2) | 32.8 (12.5)

21. Secondary Outcome: In Vivo Mitochondrial Function: QMax, VPCr
Description: Measured by 31P-mass spec. For each measure, a higher value indicates better mitochondrial function. All re calculated from multiple measures from the MRS spectra. These are relatively new research measures and normal values are not known or generally accepted.
  * QMax is theoretical maximum activity.
  * VPCr measures the rate at which PCr is regenerated.
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: mmoles/sec
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 11 | 9
mmoles/sec
  QMax | 0.42 (0.14) | 0.38 (0.13)
  VPCr | 0.24 (0.07) | 0.19 (0.08)

22. Secondary Outcome: In Vivo Mitochondrial Function: Oxidative Phosphorylation
Description: Measured by 31P-mass spec. A higher value indicates better mitochondrial function. All re calculated from multiple measures from the MRS spectra. These are relatively new research measures and normal values are not known or generally accepted. Oxidative Phosphorylation measures the rate at which electron transport activity generates phosphorylated energy sources (ATP and PCr)
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: mmol/L/s
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 11 | 9
mmol/L/s | 0.19 (0.07) | 0.13 (0.06)

23. Secondary Outcome: In Vivo Mitochondrial Function:AnGly
Description: Measured by 31P-mass spec. Anaerobic glycolysis measures the amount of anaerobic ATP generation for energy. It is generally felt that a higher value here reflects impaired mitochondrial function necessitating greater reliance on anaerobic metabolism.
Time Frame: End of each 6 week intervention period
Population: One placebo subject out of range for AnGly
Measure: Mean (Standard Deviation); unit: mmol/L/s
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 11 | 8
mmol/L/s | 0.22 (0.15) | 0.29 (0.21)

24. Secondary Outcome: Cardiac Function
Description: Cardiac output
Time Frame: End of each 6 week intervention period
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 16 | 17
L/min | 5.52 (0.76) | 4.92 (0.62)

25. Other Pre Specified Outcome: Vascular Markers: PAI-1
Description: PAI-1 exploratory thromobotic marker.
Time Frame: End of each 6 week intervention period
Population: this outcome not done-cost and assay issues
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: Vascular Markers: Exploratory
Description: ICAM
Time Frame: End of each 6 week intervention period
Population: No outcome measure data was collected for this exploratory outcome measure due to insufficient funds.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

27. Other Pre Specified Outcome: Oxidative Stress Markers
Description: TBARs, GSSG:GSH ratio
Time Frame: End of each 6 week intervention period
Population: This exploratory outcome measure was not collected
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

28. Other Pre Specified Outcome: Mitochondrial Measures: Oxidant Generation
Description: oxidant generation
Time Frame: End of each 6 week intervention period
Population: This exploratory outcome measure was not collected.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

29. Other Pre Specified Outcome: Inflammatory Markers: Exploratory
Description: IL6, TNF alpha
Time Frame: End of each 6 week intervention period
Population: No data was collected for this exploratory outcome due to insufficient funds
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

30. Other Pre Specified Outcome: Mitochondrial Oxidant Generation
Description: exploratory measure looking at H2O2 production. not performed due to equipment not available.
Time Frame: after each 6 week intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 Months
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT01813929/Prot_SAP_000.pdf